CLINICAL TRIAL: NCT01976754
Title: The Effective Dose of Dexmedetomidine for Moderate Sedation of Adult Intubated Septic Patients in the ICU.
Brief Title: Safety Study of Dexmedetomidine in Septic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, zhanqin zhang, PHD candidate, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: FirstzhejiangU
Record Dates: First submitted 2013-10-23; First posted 2013-11-06 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2016-02

CONDITIONS: Sepsis; Agitation
MeSH Terms: conditions — Sepsis; Psychomotor Agitation | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dexmedetomidine,sepsis,ED50 (Other): Intervention Name: dexmedetomidine dosage form: intravenous injection dosage：0.2-0.7μg/kg/h frequency: 1 duration:12 hours
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Septic patients are randomly received 1 of 6 doses( 0.2,0.3,0.4,0.5,0.6,0.7μg/kg/h) dexmedetomidine.
  Other Names: precedex

SUMMARY:
Septic patients in Intensive Care Unit always need mechanical ventilation and conscious-sedation. But the recommended dose 0.2-0.7μg/kg/h could not run well because of wide range. The purpose of this study is to find the effective dose of dexmedetomidine adult septic patients of mechanical ventilation .

DETAILED DESCRIPTION:
Inclusion Criteria:

Age: between 18 years mechanical ventilation RASS≥2 A diagnosis of sepsis within 48 hours

Exclusion Criteria:

Cardiac disease Cardiac rhythm abnormalities liver dysfunction coma severe hypotension muscle relaxant users

Primary Outcome Measures:

Dose of dexmedetomidine

Secondary Outcome Measures:

RASS score Requirement for rescue intervention, RASS will be recorded per hour.

ELIGIBILITY:
Inclusion Criteria:

* intubated patients RASS≥2 A diagnosis of sepsis within 48h

Exclusion Criteria:

* Cardiac disease Cardiac rhythm abnormalities liver dysfunction coma severe hypotension muscle relaxant users

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Dose of dexmedetomidine | 12 hours

SECONDARY OUTCOMES:
RASS score Requirement for rescue intervention, RASS will be recorded per hour. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: xiangming fang, PHD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- Zhanqin Zhang, Hangzhou, Zhejiang, China